CLINICAL TRIAL: NCT00048451
Title: Safety and Efficacy of Zemplar Capsule in Reducing Serum iPTH Levels in Chronic Kidney Disease Subjects (Three Times Weekly)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001-020
Record Dates: First submitted 2002-10-31; First posted 2002-11-04 (Estimated); Last update posted 2006-08-02 (Estimated); Status verified 2006-07

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — paricalcitol

INTERVENTIONS:
Drug: paricalcitol

SUMMARY:
The objective of this study is to determine whether paricalcitol is safe and effective compared to placebo in reducing elevated serum PTH levels in patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Under care of physician at least 2 months (for CKD)
* Not on active Vitamin D therapy for at least 4 weeks prior
* If female:

  * Not of childbearing potential, OR
  * Practicing birth control
  * Not breastfeeding
* If taking phosphate binders, on a stable regimen at least 4 weeks prior
* For entry into Pretreatment Phase:

  * iPTH at least 120 pg/mL
  * GFR of 15-60 mL/min and no dialysis expected for at least 6 months
* For entry into Treatment Phase:

  * Average of 2 consecutive iPTH values of at least 150 pg/mL, taken at least 1 day apart (all values not less than 120 pg/mL
  * 2 consecutive corrected serum calcium levels between 8.0-10.0 mg/dL
  * 2 consecutive serum phosphorus levels of not more than 5.2 mg/mL

Exclusion Criteria:

* History of allergic reaction or sensitivity to similar drugs
* Acute Renal Failure within 12 weeks of study
* Chronic gastrointestinal disease
* Spot urine result demonstrating a urine-calcium-to-urine creatinine ratio of greater than 0.2, or a history of renal stones
* Taken aluminum-containing phosphate binders within last 12 weeks, or requires such medication for more than 3 weeks during study
* Current malignancy, or clinically significant liver disease
* Active granulomatous disease (TB, sarcoidosis, etc.)
* History of drug or alcohol abuse within 6 mos. prior
* Evidence of poor compliance with diet or medication
* Received any investigational drug or participated in any device trial within 30 days prior
* Taking maintenance calcitonin, bisphosphonates, or drugs that may affect calcium or bone metabolism (other than females on stable estrogen and/or progestin therapy)
* On glucocorticoids for a period of more than 14 days within the last 6 months
* HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68
Dates: Start 2002-02

PRIMARY OUTCOMES:
The efficacy endpoint is achievement of two consecutive > or = 30% decreases from baseline iPTH levels.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Williams, M.D., Study Director — Abbott
Locations (19):
- United States (18):
  - Tucson Therapeutic Research Institute, Inc., Tucson, Arizona
  - Pasadena, California
  - California Institute of Renal Research, San Diego, California
  - Nephrology Educational Services and Research, Inc., Tarzana, California
  - Phoenix Internal Medicine Associates, Waterbury, Connecticut
  - University of Florida, Gainesville, Florida
  - Miami Kidney Group, Miami, Florida
  - ICSL Clinical Studies, Sarasota, Florida
  - Genesis Clinical Research Corporation, Tampa, Florida
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Medisphere Medical Research Center, Evansville, Indiana
  - Ochsner Clinic Chronic Dialysis, New Orleans, Louisiana
  - Biolab Research, LLC, Rockville, Maryland
  - The Rogosin Institute, New York, New York
  - Dialysis Clinic, Inc., Cincinnati, Ohio
  - Kidney Associates, Houston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center, San Antonio, Texas
- Wojskowy Instytut Medyczny, Warsaw, Poland